CLINICAL TRIAL: NCT02792153
Title: Estradiol and Fear Extinction for Calorie-Dense Foods in Weight Restored Adult Women With Anorexia Nervosa (AN)
Brief Title: Estradiol and Fear Extinction in Anorexia Nervosa (AN)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was withdrawn after 18 months due to lack of recruitment.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00030009
Record Dates: First submitted 2016-05-23; First posted 2016-06-07 (Estimated); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Anorexia Nervosa
Keywords: estrogen; anxiety; amenorrhea; eating disorders
MeSH Terms: conditions — Anorexia Nervosa; Anxiety Disorders; Amenorrhea; Feeding and Eating Disorders | interventions — Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Estrogen (Experimental): AN participants receive a course of transdermal estradiol treatment.
  Interventions: Drug: Estradiol

INTERVENTIONS:
Drug: Estradiol — AN participants will be prescribed 28 days of transdermal estradiol 0.1 mg/d (Days 1-28) plus 10 days (days 21-31) oral medroxyprogesterone 2.5 mg/d.
  Other Names: Climara

SUMMARY:
The purpose of this study is to determine whether estrogen may help reduce fear of high calorie-density foods in weight-restored women with Anorexia Nervosa (AN).

ELIGIBILITY:
Inclusion Criteria (AN):

* Previous diagnosis of recent AN with BMI of <18.5 (within past year)
* Current BMI > 19.0 and < 23.0 kg/m2
* Amenorrhea or oligomenorrhea

Inclusion Criteria (Healthy Controls):

* BMI > 19 < 23 kg/m2
* Taking hormone-based contraceptives for a period of one month or more
* Eating disorders symptom scores within one standard deviation of healthy controls

Exclusion Criteria (AN):

* Any medical or psychiatric problem requiring urgent medical or psychiatric attention, including acute suicidality
* History of breast cancer, deep vein thrombosis, pulmonary embolism, myocardial infarction or stroke, diabetes, liver disease, known thrombophilic disease
* Currently taking estrogen or progesterone medication
* Tobacco use greater than 1 pack per week
* Use of St. John's Wort, Phenobarbital, phenytoin, carbamazepine, rifampin, and dexamethasone can all decrease plasma estrogen level because they are CYP3A4 inducers. Cimetidine, erythromycin, clarithromycin, ketoconazole, itraconazole, ritonavir and grapefruit juice as these may increase plasma estrogen, potentially increasing the presence of side effects
* Pregnant, lactating or unwilling to use appropriate birth control (which may include abstinence) to prevent pregnancy for the duration of study participation (i.e. up to 4 weeks)
* Allergy to estradiol or medroxyprogesterone or ingredients in food items used for test meals
* Undiagnosed, abnormal vaginal bleeding

Exclusion Criteria (Healthy Controls):

* Ever diagnosed with an Eating Disorder
* Any medical or psychiatric problem requiring urgent medical or psychiatric attention, including acute suicidality
* Pregnant, lactating or unwilling to use appropriate birth control (which may include abstinence) to prevent pregnancy for the duration of study participation (i.e. up to 4 weeks)
* Food allergies to items in the test meal

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12; Primary Completion 2018-08-22 (Actual); Study Completion 2018-08-22 (Actual)

PRIMARY OUTCOMES:
Electrodermal skin conductance activity (EDA) during a test meal | Baseline (day 1) and post-treatment (day 21)
  Meal-related anxiety will be estimated from EDA recordings during a 90 minute test meal session pre- and post-treatment (day 1 and day 21). EDA will be reported as the rate of peaks (>0.02 microsiemens) per second and the average skin conductance level (in microsiemens).

SECONDARY OUTCOMES:
Heart rate variability during a test meal | Baseline (day 1) and post-treatment (day 21)
  Variability in heart rate will be measured by the variation in interpeak (beat-to-beat) interval during the 90 minute test meal session pre- and post- treatment (day 1 and day 21).
Subjective ratings of anxiety | Baseline (day 1) and post-treatment (day 21)
  Visual analog scales will be used to assess self-report anxiety at multiple points (time 0 min, 5 min, 10 min, 20 min, 30 min, 50 min, 70 min and 90 min) during the 90 minute test meal session pre- and post-treatment (day 1 and day 21).
Salivary cortisol concentration during a test meal | Baseline (day 1) and post-treatment (day 21)
  The concentration of salivary cortisol will be assessed at multiple points (time 0 min, 5 min, 10 min, 20 min, 30 min, 50 min, 70 min and 90 min) during the test meal session. Test meals occur twice during the entire length of the study on day 1 and day 21. The cortisol response will be reported as area under the curve.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Guarda, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States